CLINICAL TRIAL: NCT04453462
Title: Efficacy of Local Direct Median Nerve Block VS Brachial Plexus Block in Endoscopic Carpal Tunnel Release
Brief Title: Efficacy of Local Direct Median Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Kittipong Siriboonpipattana, Resident, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-EC-OT-6-227/61
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Carpal Tunnel Syndrome; Anesthesia, Local
Keywords: Endoscopic carpal tunnel release
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local direct median nerve block (Active Comparator): The local anesthetic technique is proposed by Wood SH and Logan AM in 1999 by using the plastic catheter to inject the anesthetic 4 cm proximally to the incision site direct over the median and ulna nerve
  Interventions: Procedure: Endoscopic carpal tunnel release under local direct median nerve block
- Brachial plexus block (Active Comparator): The brachial plexus block technique is axillary block performed under ultrasound-guided by the well-trained anesthesiologist.
  Interventions: Procedure: Endoscopic carpal tunnel release under brachial plexus block

INTERVENTIONS:
Procedure: Endoscopic carpal tunnel release under local direct median nerve block — local direct median nerve block is performed by surgeon using the 1%xylocaine with adrenaline 12 mL(5 mL subcutaneous at incision site and 7 mL over median nerve) (maximum dose 7 mg/kg) before the endoscopic carpal tunnel release(1-portal Agee technique)
  Arms: Local direct median nerve block
Procedure: Endoscopic carpal tunnel release under brachial plexus block — brachial plexus block under ultrasound-guided is performed by experienced single anesthesiologist using the 1%xylocaine with adrenaline 15 mL (maximum dose 7 mg/kg) before the endoscopic carpal tunnel release(1-portal Agee technique)
  Arms: Brachial plexus block

SUMMARY:
Carpal tunnel syndrome is the most common compressive neuropathy. Carpal tunnel release is indicated when failed conservative treatment. Although it can be done either with local anesthesia or brachial plexus block, there is no gold standard of anesthetic choice. The study is conducted to compare the efficacy of two methods and we hypothesized that the local direct median nerve block has effectiveness in intraoperative pain control not inferior to brachial plexus block in endoscopic carpal tunnel release.

DETAILED DESCRIPTION:
The study is randomized-control trial conducted in single center (Orthopaedic department, Faculty of medicine, Thammasat university) The patients with failed conservative treatment of carpal tunnel syndrome confirmed by EMG are enrolled and ramdomized with computerized block-of-4 method.The local direct median nerve block is done by the surgeon and brachial plexus block in done by single anesthesiologist after that the patient will be operated with 1-portal endoscopic carpal tunnel release (Agee technque) by single surgeon. Immediate postoperative the blinded observer will ask the patient about interaoperative pain in visual analog scale then the pateint is asked to record the 2-hr, 4-hr ,6-hr and 12-hr postoperative pain in case record form.The patient will return the case record form at 2-week and also stitched off the wound then next follow up will be 4, 12, 24 weeks to assess functional outcome (Thai version Bonton questionaire)

ELIGIBILITY:
Inclusion Criteria:

1. Patient with carpal tunnel syndrome, confirmed by EMG
2. Failed conservative treatment 3 months
3. Age ≥18 years old

Exclusion Criteria:

1. Allergic history of xylocaine
2. Any other condition that can cause carpal tunnel syndrome or peripheral neuropathy e.g. DM, hypothyroidism, pregnancy, tumor
3. Any patient that has been coverted to open carpal tunnel release

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative pain measured as visual analog scale (VAS) | Immediate postoperative period
  Visual analog scale (VAS) from 0-10 0 means no pain 5 means moderate pain 10 means worst possible pain
  Immediate postoperative the blinded observer will ask the patient about interaoperative pain in visual analog scale

SECONDARY OUTCOMES:
Postoperative pain measured as visual analog scale (VAS) | 2 hours, 4 hours, 6 hours and 12 hours postoperative period
  Visual analog scale (VAS) from 0-10 0 means no pain 5 means moderate pain 10 means worst possible pain
  The pateint is asked to record the 2 hours, 4 hours, 6 hours and 12 hours postoperative pain in case record form.
Functional outcome of the hand measured as Thai Version Boston Questionnaire | 2, 4, 12, 24 weeks postoperative period
  There are 2 parts of Thai Version Boston Questionnaire
  1. Symptom severity scores (SSS) 11 items (total score 0-55; hign score means worse outcome)
  2. Functional severity scores (FSS) 8 items (total score 0-40; hign score means worse outcome)
  The follow up will be 1, 4, 12, 24 weeks to assess functional outcome with Thai Version Boston Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chinnakart Boonyasirikool, MD, Principal Investigator — Department of Orthopaedics, Faculty of Medicine Thammasat University
Locations (1):
- Thammasat University hospital, Khlong Luang, Changwat Pathum Thani, Thailand